CLINICAL TRIAL: NCT03794037
Title: Montelukast for Prevention & Treatment of Ovarian Hyperstimulation Syndrome in Freeze-all Cycles
Brief Title: Montelukast for Prevention & Treatment of OHSS
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: no fund
Sponsor: Benha University (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Principal Investigator, Ahmed Saad, Assistant professor of Ob. & Gyn., Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Hawaa-5
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Ovarian Hyperstimulation Syndrome
Keywords: ovarian hyperstimulation syndrome; Montelukast
MeSH Terms: conditions — Ovarian Hyperstimulation Syndrome | interventions — montelukast; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): dydrgesterone 10 mg( tab)/12hs/14 days
  Interventions: Drug: dydrgesterone 10 mg( tab)/12hs/14 days
- study (Experimental): montelukast 10 mg(tab) oral/24hs/ 7 days dydrgesterone 10 mg( tab) oral/12hs/14 days
  Interventions: Combination Product: montelukast 10 mg(tab) oral/24hs/ 7 days dydrgesterone 10 mg( tab) oral/12hs/14 days

INTERVENTIONS:
Drug: dydrgesterone 10 mg( tab)/12hs/14 days — Dydrogesterone Oral Tablet 10 mg twice daily for 14 days to be taken from the day of ovum pickup
  Other Names: progesterone only
  Arms: control
Combination Product: montelukast 10 mg(tab) oral/24hs/ 7 days dydrgesterone 10 mg( tab) oral/12hs/14 days — montelukast 10 mg(tab) once daily oral for 7 days & dydrgesterone 10 mg (tab) twice daily oral for 14 days &
  Arms: study

SUMMARY:
montelukast & dydrgesteron will be given to cases with suspected or proven ovarian hyperstimulation in one group in comparison with dydrogesteron alone in the other group.

DETAILED DESCRIPTION:
patients with high risk for ovarian hyperstimulation will undergo a freeze-all protocol then montelukast & dydrgesteron will be given to cases with suspected or proven ovarian hyperstimulation in one group in comparison with dydrogesteron alone in the other group.

ELIGIBILITY:
Inclusion Criteria:

* PCOS high responders high numbers of ovum retrieved

Exclusion Criteria:

* hypersensitivity to any drug components phenylketonuria patients depression liver dysfunction

Ages: 20 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — infertile females undergoing ART cycles
Enrollment: 20 (Estimated)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants who develop ovarian hyperstimulation syndrome | 0-14 days
  incidence

SECONDARY OUTCOMES:
Number of Participants treated of ovarian hyperstimulation syndrome | 0-14 days
  treatment & resolution

CONTACTS AND LOCATIONS:
Overall Officials: ahmed sa saad, MD, ph D, Principal Investigator — Hawaa Fertility Center
Locations (1):
- Banha University- Hawaa Fertility center, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
study protocol, results,statistics
Supporting Information: Study Protocol, SAP
Time Frame: 6 months
Access Criteria: drahmedsaad@live.com